CLINICAL TRIAL: NCT01813019
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group Proof of Concept Study to Evaluate the Effect of AFQ056 in Obsessive Compulsive Disorder (OCD) Patients Resistant to Selective Serotonin Reuptake Inhibitor (SSRI) Therapy
Brief Title: Study to Evaluate the Effect of AFQ056 in Obsessive Compulsive Disorder (OCD) Patients Resistant to Selective Serotonin Reuptake Inhibitor (SSRI) Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was prematurely terminated at the time of the first Interim Analysis (IA) as the study did not meet its primary efficacy objective.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAFQ056A2225
Record Dates: First submitted 2013-03-14; First posted 2013-03-18 (Estimated); Results first posted 2016-07-21 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-11

CONDITIONS: Patient Diagnosed With OCD and Resistant to SSRI Treatment; Failed SSRI Over 12 Weeks at Appropriate Doses
Keywords: Obsessive compulsive disorder (OCD), obsessive fears, obsessions,; compulsions, OCD SSRI resistant
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Obsessive Behavior; Compulsive Behavior | interventions — mavoglurant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AFQ056 (Experimental): Following baseline, approximately 60 patients who are considered eligible will be randomized to AFQ056 arm and will receive the dosing regimen of 4 weeks AFQ056 b.i.d up-titration period of 50 mg,100 mg, 150 mg and 200 mg , followed by 12 weeks AFQ056 200 mg fixed dose* and then a 3 week down-titration of 100 mg, 50 mg and 25 mg AFQ056 b.i.d)
  *patients that do not tolerate 200 mg b.i.d may be down-titrated to 150 mg b.i.d.
  Interventions: Drug: AFQ056
- Placebo (Placebo Comparator): Following baseline, approximately 60 patients who are considered eligible will be randomized to Placebo arm and will receive the dosing regimen of 4 weeks Placebo b.i.d up-titration period of 50 mg,100 mg, 150 mg and 200 mg , followed by 12 weeks Placebo 200 mg fixed dose* and then a 3 week down-titration of 100 mg, 50 mg and 25 mg Placebo b.i.d) *patients that do not tolerate 200 matching placebo AFQ056 mg b.i.d may be down-titrated to 150 mg b.i.d.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AFQ056 — mGluR5 antagonist
  Other Names: Mavoglurant
  Arms: AFQ056
Drug: Placebo — Matched placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether AFQ056 as an add on therapy to SSRIs can have beneficial effects by reducing the total score of Y-BOCS (Yale and Brown Obsessive Compulsive Scale) in OCD patients resistant to SSRI treatment (failed SSRI over 12 weeks at appropriate doses).

DETAILED DESCRIPTION:
This was a randomized, double-blind, parallel group, placebo-controlled, 12-weeks 200 mg b.i.d oral dose treatment of AFQ056 (following a 4 week up-titration period and followed by a 3 week down-titration period) or matched placebo in patients diagnosed with OCD and on background SSRI treatment for at least 12 weeks. Study was prematurely terminated at the time of the first Interim Analysis (IA) as the study did not meet its primary efficacy objective.

ELIGIBILITY:
Inclusion Criteria:

* Male and female , non-smokers patients aged between 18 to 65 years (inclusive),
* A primary diagnosis of obsessive-compulsive disorder (OCD) as per Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-TR 4th ed, year 2000), as confirmed by an Independent Rater.
* Be on a stable appropriate dose of selective serotonin reuptake inhibitor (SSRI) treatment for at least 12 weeks prior to Baseline.
* Have an insufficient response to current SSRI treatment (as per Inclusion Criterion 4) and confirmed by an Independent Rater.
* Have a Yale-Brown Obsessive Compulsive Scale (Y-BOCS) of score ≥ 16 at Screening (and confirmed by an Independent Rater).
* Patient must have their eligibility confirmed following the remote interview conducted by the Independent Rater.
* Able to communicate well with the investigator, to understand and comply with the requirements of the study.

Exclusion Criteria:

* Diagnosis of primary OCD symptom of hoarding.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using effective methods of contraception (not including oral contraceptives) during dosing and for 30 days after last dosing of study medication.
* History of more than two unsatisfactory trials with different SSRI within a period of 2 years prior to screening (not including the current treatment with SSRI's given in an adequate dose for at least 12 weeks).
* Diagnosed with any primary DSM-IV-TR Axis I disorder other than OCD (as confirmed by an Independent Rater); with the exception of depression.
* History of eating disorder (e.g. anorexia, bulimia) according to DSMIV within the last 6 months prior to Screening, (as confirmed by an Independent Rater).
* Diagnosed with antisocial personality disorder (DSM-IV-TR Axis II), as confirmed by an Independent Rater.
* Has current or past medical history of bipolar disorder, schizophrenia or other psychotic disorders, schizoaffective disorder, autism or autistic spectrum disorders, borderline personality disorder, within the last 6 months prior to Screening.
* Smokers (use of tobacco products in the previous 3 months).
* History of hallucinations/psychosis that would require antipsychotic treatment or DSM-IV criteria being met
* Score "yes" on item 4 or item 5 of the Suicidal Ideation section of the C-SSRS, if this ideation occurred in the past 6 months, or "yes" on any item of the Suicidal Behavior section, except for the "Non- Suicidal Self-Injurious Behavior" (item also included in the Suicidal Behavior section), if this behavior occurred in the past 2 years.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (14):
- United States (3):
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Watertown, Massachusetts
  - Novartis Investigative Site, Brooklyn, New York
- Bulgaria (4):
  - Novartis Investigative Site, Burgas, Bulgaria
  - Novartis Investigative Site, Pazardzhik, Bulgaria
  - Novartis Investigative Site, Sofia, Bulgaria
  - Novartis Investigative Site, Varna, Bulgaria
- Novartis Investigative Site, Strakonice, Czech Republic, Czechia
- Germany (5):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Nuremberg
  - Novartis Investigative Site, Ulm
- Novartis Investigative Site, Bern, Switzerland

REFERENCES:
- [Derived] Rutrick D, Stein DJ, Subramanian G, Smith B, Fava M, Hasler G, Cha JH, Gasparini F, Donchev T, Ocwieja M, Johns D, Gomez-Mancilla B. Mavoglurant Augmentation in OCD Patients Resistant to Selective Serotonin Reuptake Inhibitors: A Proof-of-Concept, Randomized, Placebo-Controlled, Phase 2 Study. Adv Ther. 2017 Feb;34(2):524-541. doi: 10.1007/s12325-016-0468-5. Epub 2017 Jan 2. PMID 28044255

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Matching Placebo b.i.d. dosing
- AFQ056: AFQ056 b.i.d up-titration of 50mg,100mg, 150mg and 200 mg for 4 weeks then AFQ056 200mg b.i.d for 12 weeks and then a down-titration of AFQ056 100mg, 50mg and 25mg b.i.d for 3 weeks
Period: Overall Study
Arm/Group | Placebo | AFQ056
Started | 24 | 26
Completed | 17 | 20
Not Completed | 7 | 6
Not completed — Adverse Event | 0 | 3
Not completed — Withdrawal by Subject | 3 | 2
Not completed — administrative problems | 2 | 0
Not completed — Protocol Deviation | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | AFQ056 | Total
Number analyzed (Participants) | 24 | 26 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.9 (10.06) | 41.3 (13.27) | 40.6 (11.74)
Gender [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 11 | 13 | 24

OUTCOME MEASURES:

1. Primary Outcome: Yale - Brown Obsessive Compulsive Scale (Y-BOCS) Absolute Change From Baseline at Week 17 (End of 16-week Dosing).
Description: The Y-BOCS is a 10 item clinician-rated scale used to both determine the severity of OCD and to monitor symptom improvement throughout the course of the study. The Y-BOCS, specifically measures the severity of symptoms of OCD without being biased towards the type of obsessions or compulsions present. The scale includes questions about the amount of time spent on, how much impairment or distress experienced from, and how much resistance and control over these obsessive thoughts and compulsions. Each item is rated from 0 ("no symptoms") to 4 ("extreme symptoms") and yields a total possible score range from 0 to 40, with the following ranges indicating degree of severity:
  0-7 = sub-clinical 8-15 = mild 16-23 = moderate 24-31 = severe 32-40 = extreme Baseline was compared to week 17 (end of week 16 dosing) to produce an absolute change.
Time Frame: baseline, week 17
Population: Pharmacodynamics (PD) analysis set only participants that were analyzed at baseline and Week 17. Positive change from baseline indicates a decrease in symptom severity
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | AFQ056
Number analyzed (Participants) | 17 | 21
Scores on a scale | -8.0 (1.78) | -6.9 (1.75)
Statistical Analysis 1: Comparison: Placebo vs AFQ056; Test type: Superiority or Other; p = 0.671, Mixed Models Analysis

2. Secondary Outcome: Y-BOCS Reduction in Total Score From Baseline
Description: If a subject demonstrates at least 25% reduction in total Y-BOCS from Baseline then they will be classed as a responder whereas if a subject has a reduction in Y-BOCS of less than 25% then they will be categorized as a nonresponder.
Time Frame: 16 weeks
Population: The study was terminated due to an interim analysis of the primary efficacy outcome. Study was prematurely terminated at the time of the first Interim Analysis (IA) as the study did not meet its primary efficacy objective therefore secondary objective was not measured.
Arm/Group | Placebo | AFQ056
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Placebo | AFQ056
Serious Adverse Events (participants affected / at risk) | 2/24 | 1/26
Other Adverse Events (participants affected / at risk) | 15/24 | 18/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=24) | AFQ056 (N=26)
Atrial fibrillation (Cardiac disorders) | 1 | 0
Otitis media (Infections and infestations) | 0 | 1
Face injury (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
VIIth nerve paralysis (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=24) | AFQ056 (N=26)
Bradycardia (Cardiac disorders) | 2 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Fatigue (General disorders) | 1 | 2
Nasopharyngitis (Infections and infestations) | 4 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Disturbance in attention (Nervous system disorders) | 0 | 2
Dizziness (Nervous system disorders) | 2 | 5
Headache (Nervous system disorders) | 8 | 10
Migraine (Nervous system disorders) | 0 | 2
Abnormal dreams (Psychiatric disorders) | 1 | 2
Agitation (Psychiatric disorders) | 0 | 2
Depression (Psychiatric disorders) | 2 | 1
Insomnia (Psychiatric disorders) | 2 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.